CLINICAL TRIAL: NCT04328415
Title: Evaluation of the Blood-brain Barrier Disruption During Chronic Kidney Disease by 99mTc-DTPA Cerebral Scintigraphy (BREIN)
Brief Title: Blood-Brain Barrier Evaluation In Nephrology (BREIN)
Acronym: BREIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-42; IDRCB (Other: 2019-A02834-53)
Record Dates: First submitted 2020-03-28; First posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: End Stage Renal Disease and Cognitive Impairment
MeSH Terms: conditions — Kidney Failure, Chronic; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- healthy volunteers (Experimental)
  Interventions: Radiation: Cerebral scintigraphy
- patients with Chronic Kidney Disease (Experimental)
  Interventions: Radiation: Cerebral scintigraphy

INTERVENTIONS:
Radiation: Cerebral scintigraphy — Radioactive tracer 99mTc-DTPA

SUMMARY:
Patients with Chronic Kidney Disease (CKD) have impaired psycho-cognitive functions in parallel with deteriorating kidney function. The pathophysiology of cognitive impairment in CKD is poorly understood and there is currently no therapy to limit cognitive decline. As kidney function deteriorates, uremic toxins accumulate in the patient's body. Their cerebral toxicity, whether direct or indirect through cerebral endothelial dysfunction, is a hypothesis that may explain the cognitive abnormalities, as well as the increased severity of strokes in patients with CKD. Among uremic toxins, indoxyl sulfate (IS) is an indolic toxin that is poorly purified by dialysis and whose high levels have already been shown to be associated with an increased cardiovascular risk in patients with CKD. Our hypothesis is that the psycho-cognitive disorders observed in patients with CKD are linked to cerebral endothelial dysfunction associated with high levels of IS.

In two models of CKD in rats, found impaired cognitive performance and increased blood-brain barrier (BBB) permeability, as assessed by brain scintigraphy with 99mTc-DTPA, compared to healthy control rats. Impaired cognitive performance was correlated with BBB permeability and circulating IS levels. Rats receiving an IS-enriched diet had higher BBB permeability and more impaired cognitive performance than MRC rats without an IS-enriched diet, suggesting a central role of IS.

The 99mTc-DTPA brain scintigraphy has already been used in clinical research to assess the BBB disruption after stroke, outside the context of CKD, and the tracer is available in human nuclear medicine.

Our hypothesis is that patients with CKD would have increased permeability of the BBB compared to healthy age- and sex-matched controls, and that this permeability would correlate with circulating levels of IS as in our preclinical animal models.

The main objective of this project is to evaluate the permeability of the BBB by brain scintigraphy with 99mTc-DTPA in patients with end-stage CKD and compare it to healthy age- and sex-matched controls.

A 18-month inclusion period will allow us to recruit 15 patients with end-stage CKD and 15 healthy volunteers matched in age and gender, as an important number of patients with end-stage CKD are followed in our department. If we confirm the results obtained in animal models, we will be able to propose the analysis of BBB disruption in isotope imaging as a criterion for evaluating therapeutic approaches modulating the toxicity of indolic uremic toxins in order to limit cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* Patients :

  * over 18 years old
  * social security recipients
  * in chronic hemodialysis at least 3 times 4 hours a week for at least 3 months
  * having a negative pregnancy test less than 2 weeks old for women of childbearing age
  * who have given informed consent to participate in the study
* Healthy controls, matched in age (+/- 5 years) and sex to a patient :

  * over 18 years old
  * social security recipients
  * having a negative pregnancy test less than 2 weeks old for women of childbearing age
  * who have given informed consent to participate in the study

Exclusion Criteria:

* • Patients and healthy controls :
* Pregnant or breastfeeding women, a negative pregnancy test less than 2 weeks old will be required prior to inclusion for women of childbearing age.
* Majors under legal protection
* Lack of affiliation to a social security scheme
* Inability to give informed consent
* Persons deprived of liberty
* Date of last menstrual period > 1 month in the absence of effective contraception in patients of childbearing age with a conserved menstrual cycle
* Known neurodegenerative disease
* Major Cardiovascular Disease : Unbalanced hypertension (defined as systolic blood pressure > 160 mmHg), history of stroke or coronary artery disease.
* Ongoing neoplastic or infectious disease
* Taking non-steroidal anti-inflammatory drugs within 48 hours before inclusion
* Ongoing drug treatment that may induce attention and/or cognitive deficits (anticholinergics, sedatives, neuroleptics)
* Known hypersensitivity to the radiotracer or a component of it

  • Patients :
* Non-compliance with dialysis sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-01-07 (Estimated); Study Completion 2022-06-07 (Estimated)

PRIMARY OUTCOMES:
Ratio of intracerebral activity of 99mTc-DTPA (marker of BBB rupture) to total injected activity | 1 day
  Quantification of the intracerebral radioactivity of 99m-Tc DTPA by a senior nuclear physician, blinded from the other participants' data, in ratio to the total injected dose

CONTACTS AND LOCATIONS:
Overall Officials: Emilie GARRIDO-PRADALIE, Study Director — ASSISTANCE PUBLIQUE DES HOPITAUX DE MARSEILLE
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, France